CLINICAL TRIAL: NCT01327911
Title: A Phase 1 Multicenter Open Label Safety and Tolerability Clinical Trial of Ciliary Neurotrophic Factor (CNTF) in Patients With Macular Telangiectasia Type 2 (Mactel)
Brief Title: Ciliary Neurotrophic Factor (CNTF) Safety Trial in Patients With Macular Telangiectasia (Mactel)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Collaborators: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTMT-01
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Juxtafoveal Telangiectasia
Keywords: Mactel; Macular Telangiectasia Type 2
MeSH Terms: conditions — Idiopathic Juxtafoveal Retinal Telangiectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ciliary Neurotrophic Factor (CNTF)/NT-501 (Experimental): Biological/Vaccine:NT-501 implant
  Interventions: Biological: NT-501 implant

INTERVENTIONS:
Biological: NT-501 implant — Ciliary neurotrophic factor (CNTF) implant

SUMMARY:
This study is a phase 1, open label, non-randomized, multi-center, pilot study to evaluate the safety and tolerability of NT-501 implants in 5-7 study participants with Mactel.

DETAILED DESCRIPTION:
Protocol for Extended Follow-up of a Phase 1 Multicenter Open Label Safety and Tolerability Clinical Trial of Ciliary Neurotrophic Factor (CNTF) in Patients with Macular Telangiectasia Type 2 (MacTel)

ELIGIBILITY:
Inclusion Criteria:

* The participant must be offered sufficient opportunity to review the informed consent form, agree to the form's contents and sign the protocol's informed consent;
* The participant must have bilateral MacTel;
* Women of childbearing potential and all men must agree to use an effective form of birth control during the study;
* Participant must be medically able to undergo ophthalmic surgery for ECT implant;
* The participant's best-corrected visual acuity 64 letters or better (20/50 or better) in the study eye;

Exclusion Criteria:

* Participant is < 21 years of age;
* Participant is medically unable to comply with study procedures or follow- up visits;
* Participant has evidence of ocular disease other than MacTel that may confound the outcome of the study (e.g., diabetic retinopathy with manifest macular edema, uveitis, etc.);
* Participant has a chronic requirement (e.g., ≥ 4 weeks at a time) for ocular medications and/or has a diagnosed disease, that in the judgment of the examining physician, may be vision threatening or may affect the primary outcome (artificial tears are permitted);
* Participant has evidence of subretinal neovascularization in either eye;
* Participant has evidence of central serous chorio-retinopathy (CSR) in either eye;
* Participant has evidence of pathologic myopia in either eye;
* Participant has had a vitrectomy, penetrating keratoplasty, trabeculectomy or trabeculoplasty;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3,12, 24 and 36 months
  Visual acuity decrease of >=15 letters

SECONDARY OUTCOMES:
Microperimetry | 12, 24 and 36 months
  Change of a 10dB at least one point either adjacent to a pre-existing scotoma or in a new area within the central 10 degrees on microperimetric testing
OCT | 12, 24, and 36 months
  Change in en face area as measured by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Weng Tao, Study Chair — Neurotech USA
Locations (2):
- United States (2):
  - Jules Stein Eye Institute, Los Angeles, California
  - Retina Associates of Cleveland, Cleveland, Ohio